CLINICAL TRIAL: NCT06767033
Title: Inferior Vena Cava Collapsibility Index Assessment in Predicting Post Spinal Anaesthesia Hypotension in Patients Undergoing Arthroscopic Knee Surgeries.
Status: Completed | Type: Observational
Sponsor: Ain Shams University (Other)
Responsible Party: Sponsor
Other Study IDs: FMASU MS89/2024
Record Dates: First submitted 2025-01-05; First posted 2025-01-09 (Actual); Last update posted 2025-01-09 (Actual); Status verified 2024-09

CONDITIONS: Post Spinal Anaesthesia Hypotension; Inferior Vena Cava Collapsibility Index
Keywords: Inferior Vena Cava Collapsibility Index; Post Spinal Anaesthesia Hypotension; Arthroscopic Knee Surgeries

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

INTERVENTIONS:
Device: Ultrasound Guided Inferior Vena Cava Collapsibility Index Assessment — Before spinal anaesthesia, inferior vena cava collapsibility index was measured for all patients using Ultrasound device.

SUMMARY:
The aim of this study was to evaluate the role of inferior vena cava collapsibility index assessment in predicting post spinal anaesthesia hypotension in patients undergoing arthroscopic knee surgeries.

DETAILED DESCRIPTION:
Prospective Cohort Study conducted in Ain Shams University Hospitals.

ELIGIBILITY:
Inclusion Criteria:

* Patients: American Society of Anesthesiologists Physical Status (ASA) I to II undergoing arthroscopic knee surgeries under spinal anaesthesia.
* Both Sexes.
* Aged 30 to 60 years.
* Body mass index <35 kg/m2

Exclusion Criteria:

* Patients' refusal of procedure or participation in the study.
* Patients with contraindication to spinal anaesthesia.
* Patients with severe cardiovascular or pulmonary disease.
* Patients with pre-procedural hypotension (systolic arterial pressure less than 90 mmHg and/or mean arterial pressure less than 60 mmHg).

Ages: 30 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Patients American Society of Anesthesiologists Physical Status (ASA) I to II undergoing arthroscopic knee surgeries under spinal anaesthesia.
Sampling Method: Non-Probability Sample
Enrollment: 40 (Actual)
Dates: Start 2024-02-22 (Actual); Primary Completion 2024-08-22 (Actual); Study Completion 2024-09-01 (Actual)

PRIMARY OUTCOMES:
to determine the optimal cut-off value of ultrasound guided IVCCI to predict post spinal anaesthesia hypotension. | 6 months

SECONDARY OUTCOMES:
to measure the total amount of fluids and vasopressor drugs administered to patients to manage post spinal anaesthesia hypotension | 6 months

CONTACTS AND LOCATIONS:
Locations (1):
- Ain Shams University Hospitals, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: Undecided